CLINICAL TRIAL: NCT04032444
Title: Collecting Orthopedic Safety and Performance Data Using Surgeons Clinical Outcomes Registry (SCOR)
Acronym: SCOR
Status: Terminated | Type: Observational
Why Stopped: Sponsor terminated. No longer needed to support business need
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: 19F-W-SCOR-RM
Record Dates: First submitted 2019-07-16; First posted 2019-07-25 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Orthopedics
Keywords: Orthopedic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Surgeons Clinical Outcomes Registry (SCOR) is a global registry designed to collect safety and performance data on commercially available Wright Medical products. Registry data may be used for publications, education and marketing materials, post-market surveillance, future regulatory submissions, research and development for product design, software improvements, and development of artificial intelligence learning and tools.

ELIGIBILITY:
Inclusion criteria:

• Patients 18 years of age or older that have or will be receiving a Wright Medical product

Exclusion criteria:

• Member of a vulnerable population, including minors, those unable to decide for themselves to participate or needing a Legally Authorized Representative (LAR), or others who could be subject to coercion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from United States, Europe, Canada and Australia.
Sampling Method: Non-Probability Sample
Enrollment: 723 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Number of device associated and procedure associated adverse events. | up to 20 years

SECONDARY OUTCOMES:
Rates of revision surgeries. | up to 20 years

OTHER OUTCOMES:
Time to first revision surgery. | up to 20 years
Change from baseline to previous visit in ASES scores | Standard of care follow up visits up to 20 years
  ASES Score = American Shoulder and Elbow Surgeons Score, 11 items with total score reported out of 100 measuring pain and activity of patient's evaluated shoulder where lower scores indicate more pain and less function
Change from baseline to previous visit in Constant Murley scores | Standard of care follow up visits up to 20 years
  Combination of physician-completed and patient-reported portions to assess functional state of shoulder including range of motion; total score reported out of 100 measuring where lower scores indicate less function of the evaluated shoulder
Change from baseline to previous visit in SANE scores | Standard of care follow up visits up to 20 years
  SANE = Single Assessment Numeric Evaluation; 1 item assessment of shoulder rating 0% to 100%
Change from baseline to previous visit in Patient Satisfaction scores | Standard of care follow up visits up to 20 years
  Single, subjective question measuring patient satisfaction; assessed by improved, worsened, or no change in satisfaction
Change from baseline to previous visit in SST scores | Standard of care follow up visits up to 20 years
  SST = Simple Shoulder Test; 12 Y/N questions assessing patient's perspective of shoulder function scored out of 100% where lower scores indicate less function
Change from baseline to previous visit in WOOS scores | Standard of care follow up visits up to 20 years
  WOOS = Western Ontario Osteoarthritis of the Shoulder; 19 items measuring quality of life specific to patient's shoulder. Each item is out of 100, where a total score is summed where the worst possible score is 1900, the aggregate score is subtracted from 1900 and divided by 19 to provide the score in a % out of 100% with 100% being worst score.
Change from baseline to previous visit in PROMIS scores | Standard of care follow up visits up to 20 years
  PROMIS Global Health = Patient-Reported Outcomes Measurement Information System - Global Health questionnaire; The PROMIS Global-10 is a 10-item patient-reported questionnaire in which the response options are presented as 5-point (as well as a single 11-point) rating scales. Higher scores indicate a healthier patient with a total score of 50.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Chaoui, PhD, MSc, Principal Investigator — Stryker Trauma and Extremities
Locations (7):
- United States (7):
  - Orthopedic Surgeon, Bradenton, Florida
  - Orthopedic Surgeon, Augusta, Georgia
  - Orthopedic Surgeon, Orland Park, Illinois
  - Orthopedic Surgeon, Indianapolis, Indiana
  - Orthopedic Surgeon, Peabody, Massachusetts
  - Orthopedic Surgeon, Florham Park, New Jersey
  - Orthopedic Surgeon, Woodbridge, Virginia